CLINICAL TRIAL: NCT04616677
Title: An Open-Label, Single-Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-42847922 in Adult Participants.
Brief Title: A Study to Evaluate the Effect of Renal Impairment on JNJ-42847922 in Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108903; 42847922MDD1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Parts 1 and 2: Cohort 1 (JNJ-42847922) (Active Comparator): Healthy participants with normal renal function [estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter (mL)/minute (min)] will receive single oral dose of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 1: Cohort 2 (JNJ-42847922) (Experimental): Participants with severe renal impairment (eGFR 15 to 29 mL/min) will receive single oral dose of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 2 (Optional): Cohort 3 (JNJ-42847922) (Experimental): Participants with moderate renal impairment (eGFR 30 to 59 mL/min) will receive single oral dose of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922

INTERVENTIONS:
Drug: JNJ-42847922 — JNJ-42847922 tablet will be administered orally.
  Other Names: Seltorexant

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic of a single oral dose of JNJ-42847922 in adult participants with renal impairment compared with healthy participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kilogram {kg}]/height [meter {m}]^2) between 18 and 40 kilograms per meter square (kg/m^2) (inclusive) with a body weight not less than 50 kg
* All female participants (regardless of childbearing potential), must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day 1
* Must not donate blood for up to 3 months after study
* Participants with normal renal function (Group 1) must meet the following additional inclusion criteria to be enrolled in the study: Must have normal renal function defined as: estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter (mL)/minute (min) at screening
* Participants with moderate (optional Group 3) or severe (Group 2) renal impairment must meet the following additional inclusion criteria to be enrolled in the study: Must have a eGFR of less than (<) 90 mL/min with the following classification used at screening: Moderate renal impairment (eGFR >= 30 to 59 mL/min); Severe renal impairment (eGFR >= 15 to 29 mL/min)
* Participants with moderate (optional Group 3) or severe (Group 2) renal impairment must meet the following additional inclusion criteria to be enrolled in the study: Must have stable renal function, that is, no significant change in renal function as evidenced by the (mean) screening serum creatinine value within plus minus (+ -) 25 percent (%) from the determination obtained at least 3 months prior to screening, and expected to remain stable during the study, and not planning to initiate dialysis

Exclusion Criteria:

* Participants who: are on a vegetarian diet or who take creatine supplements, have a non-standard muscle mass, such as, amputation, malnutrition, or muscle wasting, because these factors are not accounted for in the prediction equations for glomerular filtration rate (GFR)
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 5 times the drug's half-life, whichever is longer, before study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Participants with renal impairment (Cohort 2 and Cohort 3) have kidney failure, requiring dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-42847922 and its Metabolites A and B | Pre-dose, up to 96 hours post-dose (up to Day 5)
  Cmax is defined as maximum observed plasma analyte concentration of JNJ-42847922 and its metabolites A and B.
Area Under Plasma Analyte Concentration versus Time Curve from Time 0 to Time of Last Measurable Concentration (AUC [0-Last]) of JNJ-42847922 and its Metabolites A and B | Pre-dose, up to 96 hours post-dose (up to Day 5)
  AUC(0-Last) is defined as area under the plasma analyte concentration versus time curve from time 0 to time of last measurable concentration of JNJ-42847922 and its metabolites A and B.
Area Under the Plasma Analyte Concentration versus Time Curve from Time 0 to Infinite Time (AUC[0-Infinity]) of JNJ-42847922 and its Metabolites A and B | Pre-dose, up to 96 hours post-dose (up to Day 5)
  AUC(0-infinity) is defined as the area under the plasma analyte concentration versus time curve from time 0 to infinite time of JNJ-42847922 and its metabolites A and B.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 5
  An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency